CLINICAL TRIAL: NCT04111666
Title: A Phase 1 Study in Healthy Volunteers to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Bioavailability of IV and SC AL101
Brief Title: A Phase 1 First in Human Study to Assess Safety and Tolerability of AL101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL101-1
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AL101 IV (Experimental): * Up to four single ascending doses (SAD IV cohorts)
  * Multiple doses of AL101 administered IV (MD IV cohort)
  Interventions: Biological: AL101
- Saline Solution (Placebo Comparator): Saline solution will be administered with the following:
  * Single IV infusion for four single ascending doses (SAD IV cohorts) in a ratio of 8 active and 3 placebo subjects
  * Multiple IV infusions for the MD IV cohort in a ratio of 8 active and 2 placebo subjects
  Interventions: Other: Placebo
- AL101 SC (Experimental): * Single fixed dose levels of AL101 administered SC
  * Multiple fixed dose of AL101 administered SC
  Interventions: Biological: AL101

INTERVENTIONS:
Biological: AL101 — Active dose of AL101
  Arms: AL101 IV; AL101 SC
Other: Placebo — Saline solution administered as a single and multiple infusion as placebo.
  Arms: Saline Solution

SUMMARY:
A first in human phase 1 study in healthy volunteers to assess AL101 safety, tolerability, bioavailability, pharmacokinetics, and pharmacodynamics

DETAILED DESCRIPTION:
This is a first-in-human Phase 1 study designed to investigate the safety, tolerability, PK, PD and Bioavailability of intravenously and sub-cutaneously administered AL101 in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.0-35.0 kg/m2
* 45-120 kg, inclusive
* At screening, females must be non-pregnant and non-lactating, or of nonchildbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1-year postmenopausal (amenorrhoea duration of 12 consecutive months); nonpregnancy will be confirmed for all females by a pregnancy test conducted at screening, (each) admission, and at follow-up.
* Female participants of child-bearing potential must agree to use adequate contraception from screening until 90 days after the follow-up visit.
* In good physical health on the basis of no clinically significant findings from medical history, physical examination (PE), laboratory tests, 12 lead ECG, and vital signs, as judged by the Investigator.
* Willingness and able to comply with the study protocol, in the investigator's judgement.

Exclusion Criteria:

* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Positive drug or alcohol at screening and prior to first dose
* History of alcohol abuse or substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of AL101 measured by number of subjects with adverse events and Dose Limiting Adverse Event (DLAEs) | either 57, 113, or 141 days, depending on the cohort
  Incidence of adverse events and dose limiting Adverse Events during the DLAE observation period and/or study treatment periods.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AL101 | either 57, 113, or 141 days, depending on the cohort
  Serum and CSF concentration of AL101 at specified time points
Maximum plasma concentration (Cmax) for AL101 | either 57, 113, or 141 days, depending on the cohort
  Evaluate Cmax for serum and CSF concentration of AL101 at specified time points
Area under the curve concentration (AUC) for AL101 | either 57, 113, or 141 days, depending on the cohort
  Evaluate AUC for serum and CSF concentration of AL101 at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Kusnir, Principal Investigator — Bioclinica Research; Maria Bermudez, Principal Investigator — Quotient Sciences
Locations (2):
- United States (2):
  - Study site, Miami, Florida
  - Study site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budda B, Mitra A, Park L, Long H, Kurnellas M, Bien-Ly N, Estacio W, Burgess B, Chao G, Schwabe T, Paul R, Kenkare-Mitra S, Rosenthal A. Development of AL101 (GSK4527226), a progranulin-elevating monoclonal antibody, as a potential treatment for Alzheimer's disease. Alzheimers Res Ther. 2025 Jul 25;17(1):174. doi: 10.1186/s13195-025-01817-4. PMID 40713730